CLINICAL TRIAL: NCT01076738
Title: The Value of Routine Screening for Diffuse Vascular Disease in the Canadian Post-Acute Coronary Syndrome/Ischemic Stroke/Transient Ischemic Attack General Practice Population With Previously Undocumented Peripheral Arterial Disease
Brief Title: Screening DIVA - Diffuse Vascular Disease
Status: Completed | Type: Observational
Sponsor: Sanofi (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Medical Affairs study director, sanofi-aventis
Other Study IDs: DIREG_L_04222
Record Dates: First submitted 2010-02-25; First posted 2010-02-26 (Estimated); Last update posted 2010-09-13 (Estimated); Status verified 2010-09

CONDITIONS: Peripheral Vascular Diseases
MeSH Terms: conditions — Peripheral Vascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- single group study

SUMMARY:
Primary Objective:

To investigate the value of the Edinburgh Claudication Questionnaire (ECQ) against the ankle-brachial index (ABI) in Canadian patients mainly followed in general practice, with documented acute coronary syndrome (ACS)/ischemic stroke (IS)/transient ischemic attack (TIA) and who are not known to have peripheral arterial disease (PAD) at the time of enrolment.

Secondary Objective:

To collect data on the prevalence of PAD in this population as measured by ABI.

ELIGIBILITY:
Inclusion Criteria:

* Documented acute coronary syndrome (Unstable angina, non-Q-wave myocardial infarction, Q-wave myocardial infarction) or/and documented ischemic stroke/transient ischemic attack (IS/TIA)

Exclusion Criteria:

* Previously known symptomatic or asymptomatic PAD confirmed by one of the following diagnostic methods or interventions (documented in the patient's medical record):

  * Non-invasive or invasive vascular diagnostic tools (e.g.: ABI, Toe-brachial index, Duplex ultrasound, Magnetic resonance angiography, Computer tomographic angiography, Contrast angiography)
  * Previous related intervention (such as angioplasty, stenting, atherectomy, peripheral arterial bypass graft, other vascular intervention including amputation)
* Patients whose ABI cannot be measured accurately
* Patients already in a clinical trial or a product registry
* Hospitalized patients

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with documented ACS or/and IS / TIA
Sampling Method: Non-Probability Sample
Enrollment: 2233 (Estimated)
Dates: Start 2009-04; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
To determine the sensitivity and specificity of the ECQ versus ABI. | within 12 (+/- 2) weeks

SECONDARY OUTCOMES:
To determine the prevalence of symptomatic PAD (positive ECQ and ABIT <0.9) | within 12 (+/- 2) weeks
To determine the prevalence of asymptomatic PAD (negative ECQ and ABI <0.9) | within 12 (+/- 2) weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Affairs, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Laval, Canada

REFERENCES:
- [Derived] Bell AD, Roussin A, Popovici-Toma D, Girard M, Chiu JF, Huckell V. The value of routine screening for peripheral arterial disease in stable outpatients with a history of coronary artery or cerebrovascular disease. Int J Clin Pract. 2013 Oct;67(10):996-1004. doi: 10.1111/ijcp.12148. Epub 2013 May 21. PMID 23692499